CLINICAL TRIAL: NCT03289728
Title: Evaluation of a Strategy Guided by Imaging Versus Systematic Coronary Angiography in Elderly Patients With Ischemia: a Multicentric Randomized Non Inferiority Trial.
Brief Title: Evaluation of a Strategy Guided by Imaging Versus Systematic Coronary Angiography in Elderly Patients With Ischemia
Acronym: EVAOLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.012
Record Dates: First submitted 2017-06-07; First posted 2017-09-21 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Infarction
Keywords: elderly patients; myocardial infarction; myocardial revascularization strategy; ischemia imaging; coronary artery disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy guided by ischemia imaging (Experimental): Non-invasive imaging (SPECT or DSE) will be performed. High-risk Patients judged to high risk by imaging (according to ESC guidelines (5)) will undergo coronary angiography aimed at myocardial revascularization and have optimal medical treatment, according to ESC guidelines.
  - Low or intermediate risk patients will receive optimal medical treatment.
  Interventions: Other: Stress single photon emission CT (SPECT) or Stress ultrasound with dobutamine (DSE)
- Systematic coronary angioplasty (Active Comparator): Patients will routinely undergo invasive coronary angiography aimed at myocardial revascularization.
  Interventions: Procedure: Cornorary angioplasty

INTERVENTIONS:
Other: Stress single photon emission CT (SPECT) or Stress ultrasound with dobutamine (DSE) — Stress single photon emission CT (SPECT) or Stress ultrasound with dobutamine (DSE), performed using standard protocol.
  Patients with ≥ moderate ischemia observed by SPECT (≥ 10% of the myocardium or transient ischaemic dilatation or reduced post-stress ejection fraction (EF)) or abnormal movements of the myocardial walls observed during a stress echocardiogram (≥ 3/17 segments) will benefit from coronary angiography. Depending on the results of coronary angiography and on the coronary anatomy and other clinical and para-clinical considerations (territory of myocardial ischemia) revascularisation will be performed (REVASC). Patients with < moderate ischemia will receive medical treatment only (MT).
  Arms: Strategy guided by ischemia imaging
Procedure: Cornorary angioplasty — Participants randomized to the SCA group, will benefit from a coronary angiography within 24 to 72 hours after the diagnosis of NSTEMI; without any preliminary ischemia imaging.
  Arms: Systematic coronary angioplasty

SUMMARY:
The WHO predicts that cardiovascular morbi-mortality will increase by 120-137% within 20 years due to the aging population. Myocardial infarction without ST segment elevation (NSTEMI) is the most common form of infarction. However, its treatment among elderly patients remains a challenging question.

Indeed, the risk benefit balance of revascularization remains unclear, and complications related to revascularization are more frequent in the elderly, including MI, heart failure, stroke, renal failure and bleeding according to National Cardiovascular Network data.The last randomized controlled trial "After Eighty Study", showed a reduction of major cardio-cerebrovascular events (MACCEs) in NSTEMI patients with an invasive strategy (systematic coronary angiography - CA) compared to a conservative strategy (medical treatment alone). Nevertheless, this study presented several limitations of which a major one was the lack of a definition of frailty at inclusion. Moreover, the "After Eighty Study" has shown that percutaneous revascularization in the invasive arm was only performed for 1 in 2 patients showing an inadequacy in the strategy for selecting candidates for revascularization.

Consequently, despite European Society of Cardiology (ESC) guidelines, the management of NSTEMI in elderly patients is not yet evidence based, and current recommendations do not provide any clear clinical decision rule indicating one strategy over another.

For fragile patients, an alternative strategy consists of selecting candidates for a guided CA according to the extent of myocardial ischemia, identified by non-invasive imaging. Single-photon emission computed tomography or dobutamine stress echocardiograms are currently the reference methods with well-defined interpretation of ischemia. According to our experience, this strategy avoids CA for one third of patients and improves the rate of revascularization.

The aim of our study is to compare 1-year morbidity and mortality in NSTEMI patients over 80 years, assigned to guided versus systematic-CA. Our hypothesis is that the guided strategy will not be inferior on MACE rates at 1 year, and will be cost-effective by reducing iatrogenic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 80 years or older
* Hospitalized for NSTEMI with or without ST-segment depression on electrocardiogram (ECG), and with raised blood concentration of troponin T or I. Raised troponin was defined as a value exceeding the 99th percentile of a normal population at the local laboratory at each participating site. A local cardiologist assessed patient eligibility and clinical condition compatible with a doubt for systematic coronary angiography due to a frailty.
* Written informed consent by the patient or the next of kin in case of incapacity.

Non-inclusion criteria:

* Recurrent or ongoing chest pain refractory to medical treatment
* Haemodynamic instability or cardiogenic shock
* Life-threatening arrhythmias or cardiac arrest
* Contra-indication to CA: Renal failure (creatinine clearance <15 mL/min by Modification of the Diet in Renal Disease (MDRD)), continuing bleeding problems
* Mechanical complications of MI
* Severe aortic stenosis
* Medical history of severe dementia (documented for more than 3 months)
* Patient under administrative or judicial control
* Patient who are protected under the act
* No health care insurance

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1756 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of MACCE | 12 months
  Rate of MACCE (defined as all-cause death, non-fatal myocardial infarction, non-fatal stroke)

SECONDARY OUTCOMES:
Rate of MACCEs and each component of the MACCEs criteria during index hospitalization | 1, 6 and 12 months
  MACCE (defined as all-cause death, non-fatal myocardial infarction, non-fatal stroke)
Incremental cost-effectiveness ratio (ICER) expressed as the extra cost for a QALY (quality adjusted life year) gained by the strategy guided by ischemia imaging compared to the systemic coronary angioplasty strategy | 12 months
The annual financial impact of implementing the strategy guided by ischemia imaging will be calculated from the French Health Insurance System perspective over three years | 12 months
Quality of life using standardized scale : EQ5D-5L | 1, 6 and 12 months
Frailty assessment | 1 week
  Multiple assessment are necessary to evaluate patient frailty: ADL, IADL, CAM, MNA, Charlson score, SEGA, MMSE, Time up and go test, mini GDS, history of fall
Dependency (ADL) | 1, 6, 12 months
Autonomy (IADL) | 1, 6, 12 months
Incidence of bledding events as defined by the Bleeding Research Consortium (BARC) score ≥ 3 | 1. 6, 12 months
Rate of MACCE according to sub-group analysis | 1. 6, 12 months
  Sub group : age, gender, diabetes, renal failure and frailty
Create prognostic model with multivariate survival analysis : | 1. 6, 12 months
  Risk Algorithm, setting up a score to choose an invasive strategy or not based on analysis of different score (for example geriatric score)
Rate of all-cause death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, resuscitated cardiac arrest and ischemia-driven coronary revascularization procedure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Barone-Rochette, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Clinique Mutualiste, Grenoble
  - University Hospital Grenoble, Grenoble

REFERENCES:
- [Result] Batchelor WB, Anstrom KJ, Muhlbaier LH, Grosswald R, Weintraub WS, O'Neill WW, Peterson ED. Contemporary outcome trends in the elderly undergoing percutaneous coronary interventions: results in 7,472 octogenarians. National Cardiovascular Network Collaboration. J Am Coll Cardiol. 2000 Sep;36(3):723-30. doi: 10.1016/s0735-1097(00)00777-4. PMID 10987591
- [Result] Bauer T, Koeth O, Junger C, Heer T, Wienbergen H, Gitt A, Zahn R, Senges J, Zeymer U; Acute Coronary Syndromes Registry (ACOS) Investigators. Effect of an invasive strategy on in-hospital outcome in elderly patients with non-ST-elevation myocardial infarction. Eur Heart J. 2007 Dec;28(23):2873-8. doi: 10.1093/eurheartj/ehm464. Epub 2007 Nov 2. PMID 17982163
- [Result] Rosengren A, Wallentin L, Simoons M, Gitt AK, Behar S, Battler A, Hasdai D. Age, clinical presentation, and outcome of acute coronary syndromes in the Euroheart acute coronary syndrome survey. Eur Heart J. 2006 Apr;27(7):789-95. doi: 10.1093/eurheartj/ehi774. Epub 2006 Feb 7. PMID 16464911
- [Result] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Result] Alexander KP, Anstrom KJ, Muhlbaier LH, Grosswald RD, Smith PK, Jones RH, Peterson ED. Outcomes of cardiac surgery in patients > or = 80 years: results from the National Cardiovascular Network. J Am Coll Cardiol. 2000 Mar 1;35(3):731-8. doi: 10.1016/s0735-1097(99)00606-3. PMID 10716477
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Wallentin L, Lagerqvist B, Husted S, Kontny F, Stahle E, Swahn E. Outcome at 1 year after an invasive compared with a non-invasive strategy in unstable coronary-artery disease: the FRISC II invasive randomised trial. FRISC II Investigators. Fast Revascularisation during Instability in Coronary artery disease. Lancet. 2000 Jul 1;356(9223):9-16. doi: 10.1016/s0140-6736(00)02427-2. PMID 10892758
- [Result] Lagerqvist B, Husted S, Kontny F, Stahle E, Swahn E, Wallentin L; Fast Revascularisation during InStability in Coronary artery disease (FRISC-II) Investigators. 5-year outcomes in the FRISC-II randomised trial of an invasive versus a non-invasive strategy in non-ST-elevation acute coronary syndrome: a follow-up study. Lancet. 2006 Sep 16;368(9540):998-1004. doi: 10.1016/S0140-6736(06)69416-6. PMID 16980115
- [Result] Fox KA, Clayton TC, Damman P, Pocock SJ, de Winter RJ, Tijssen JG, Lagerqvist B, Wallentin L; FIR Collaboration. Long-term outcome of a routine versus selective invasive strategy in patients with non-ST-segment elevation acute coronary syndrome a meta-analysis of individual patient data. J Am Coll Cardiol. 2010 Jun 1;55(22):2435-45. doi: 10.1016/j.jacc.2010.03.007. Epub 2010 Mar 30. PMID 20359842
- [Result] Savonitto S, Cavallini C, Petronio AS, Murena E, Antonicelli R, Sacco A, Steffenino G, Bonechi F, Mossuti E, Manari A, Tolaro S, Toso A, Daniotti A, Piscione F, Morici N, Cesana BM, Jori MC, De Servi S; Italian Elderly ACS Trial Investigators. Early aggressive versus initially conservative treatment in elderly patients with non-ST-segment elevation acute coronary syndrome: a randomized controlled trial. JACC Cardiovasc Interv. 2012 Sep;5(9):906-16. doi: 10.1016/j.jcin.2012.06.008. PMID 22995877
- [Result] Tegn N, Abdelnoor M, Aaberge L, Endresen K, Smith P, Aakhus S, Gjertsen E, Dahl-Hofseth O, Ranhoff AH, Gullestad L, Bendz B; After Eighty study investigators. Invasive versus conservative strategy in patients aged 80 years or older with non-ST-elevation myocardial infarction or unstable angina pectoris (After Eighty study): an open-label randomised controlled trial. Lancet. 2016 Mar 12;387(10023):1057-1065. doi: 10.1016/S0140-6736(15)01166-6. Epub 2016 Jan 13. PMID 26794722
- [Result] Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. 2014 Mar 4;63(8):747-62. doi: 10.1016/j.jacc.2013.09.070. Epub 2013 Nov 27. PMID 24291279
- [Result] Ekerstad N, Swahn E, Janzon M, Alfredsson J, Lofmark R, Lindenberger M, Carlsson P. Frailty is independently associated with short-term outcomes for elderly patients with non-ST-segment elevation myocardial infarction. Circulation. 2011 Nov 29;124(22):2397-404. doi: 10.1161/CIRCULATIONAHA.111.025452. Epub 2011 Nov 7. PMID 22064593
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S. [2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC)]. G Ital Cardiol (Rome). 2016 Oct;17(10):831-872. doi: 10.1714/2464.25804. No abstract available. Italian. PMID 27869901
- [Result] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Result] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. J Am Coll Cardiol. 2007 Nov 27;50(22):2173-95. doi: 10.1016/j.jacc.2007.09.011. No abstract available. PMID 18036459
- [Result] Manrique A, Marie PY, Agostini D, Maunoury C, Acar P; Groupe de travail Cardiologie nucleaire et IRM. [Update of recommendations for nuclear cardiology stress tests in adults and children]. Arch Mal Coeur Vaiss. 2002 Sep;95(9):851-72. No abstract available. French. PMID 12407803
- [Result] Furber A, Berdague P, Cadiou C, David N, Faraggi M, Fourquet N, Helias J, Le Guludec D, Marie PY, Ouhayoun E, Pezard P, Vanzetto G, Weinmann P; Groupe de travail Cardiologie nucleaire et IRM. [Recommendations of the French Society of Cardiology concerning the practice of ischemia provocation tests in adult nuclear cardiology]. Arch Mal Coeur Vaiss. 2000 Nov;93(11):1309-32. No abstract available. French. PMID 11190460
- [Result] Manrique A, Marie PY; Nuclear Cardiology MRI Group. [Recommendations for the performance and interpretation of myocardial perfusion tomoscintigraphy]. Arch Mal Coeur Vaiss. 2003 Jun;96(6):695-711. No abstract available. French. PMID 12868353
- [Result] Verberne HJ, Acampa W, Anagnostopoulos C, Ballinger J, Bengel F, De Bondt P, Buechel RR, Cuocolo A, van Eck-Smit BL, Flotats A, Hacker M, Hindorf C, Kaufmann PA, Lindner O, Ljungberg M, Lonsdale M, Manrique A, Minarik D, Scholte AJ, Slart RH, Tragardh E, de Wit TC, Hesse B; European Association of Nuclear Medicine (EANM). EANM procedural guidelines for radionuclide myocardial perfusion imaging with SPECT and SPECT/CT: 2015 revision. Eur J Nucl Med Mol Imaging. 2015 Nov;42(12):1929-40. doi: 10.1007/s00259-015-3139-x. Epub 2015 Aug 21. PMID 26290421
- [Result] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Int J Cardiovasc Imaging. 2002 Feb;18(1):539-42. No abstract available. PMID 12135124
- [Result] Sicari R, Nihoyannopoulos P, Evangelista A, Kasprzak J, Lancellotti P, Poldermans D, Voigt JU, Zamorano JL; European Association of Echocardiography. Stress Echocardiography Expert Consensus Statement--Executive Summary: European Association of Echocardiography (EAE) (a registered branch of the ESC). Eur Heart J. 2009 Feb;30(3):278-89. doi: 10.1093/eurheartj/ehn492. Epub 2008 Nov 11. No abstract available. PMID 19001473
- [Result] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Result] Lakatos E, Lan KK. A comparison of sample size methods for the logrank statistic. Stat Med. 1992 Jan 30;11(2):179-91. doi: 10.1002/sim.4780110205. PMID 1579757
- [Result] Com-Nougue C, Rodary C, Patte C. How to establish equivalence when data are censored: a randomized trial of treatments for B non-Hodgkin lymphoma. Stat Med. 1993 Jul 30;12(14):1353-64. doi: 10.1002/sim.4780121407. PMID 8210831
- [Result] Rothmann M, Li N, Chen G, Chi GY, Temple R, Tsou HH. Design and analysis of non-inferiority mortality trials in oncology. Stat Med. 2003 Jan 30;22(2):239-64. doi: 10.1002/sim.1400. PMID 12520560
- [Result] Fleming TR, Harrington DP, O'Brien PC. Designs for group sequential tests. Control Clin Trials. 1984 Dec;5(4):348-61. doi: 10.1016/s0197-2456(84)80014-8. PMID 6518769
- [Result] Chevalier J, de Pouvourville G. Valuing EQ-5D using time trade-off in France. Eur J Health Econ. 2013 Feb;14(1):57-66. doi: 10.1007/s10198-011-0351-x. Epub 2011 Sep 21. PMID 21935715
- [Result] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198
- [Result] Sullivan SD, Mauskopf JA, Augustovski F, Jaime Caro J, Lee KM, Minchin M, Orlewska E, Penna P, Rodriguez Barrios JM, Shau WY. Budget impact analysis-principles of good practice: report of the ISPOR 2012 Budget Impact Analysis Good Practice II Task Force. Value Health. 2014 Jan-Feb;17(1):5-14. doi: 10.1016/j.jval.2013.08.2291. Epub 2013 Dec 13. PMID 24438712
- [Derived] Barone-Rochette G, Vanzetto G, Danchin N, Steg PG, Hanon O, Charlon C, David-Tchouda S, Gavazzi G, Simon T, Bosson JL; EVAOLD study investigator. Rationale and design of the multicentric randomized EVAOLD trial: Evaluation of a strategy guided by imaging versus routine invasive strategy in elderly patients with ischemia. Am Heart J. 2025 Jan;279:94-103. doi: 10.1016/j.ahj.2024.10.013. Epub 2024 Oct 23. PMID 39447717